CLINICAL TRIAL: NCT03629782
Title: Characterisation of Patients With Severe Asthma in Primary and Secondary Care Settings in Europe Reported to be Eligible for Biological Therapy
Acronym: RECOGNISE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00039
Record Dates: First submitted 2018-04-24; First posted 2018-08-14 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-country, multicentre, observational cross-sectional one-visit study of patients suffering from severe asthma in primary and secondary care settings in Europe

DETAILED DESCRIPTION:
This study aims to generate real-world data on the characteristics of patients considered to have severe asthma in primary and secondary care settings that should be referred for assessment for biologics. It is anticipated that these data from European countries, will help to estimate the unmet need for better treatments in severe asthma patients and will provide supporting evidence on the current shortcomings in referrals to asthma specialist or secondary care clinics. This information could also support the development of better severe asthma care pathways across Europe.

Approximately 1,500 other patients like you will take part in the RECOGNISE study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older with physician's confirmed diagnosis of asthma.
* Diagnosis of asthma defined as severe according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines, i.e.: Asthma requiring high-dose ICS plus at least one of the following additional controller[s] for 12 months (GINA Step 4/5): Long-acting beta2-agonist (LABA), leukotriene modifier, theophylline, or continuous or near continuous OCS [i.e.,maintenance OCS for ≥50% of the previous year])(controlled or uncontrolled). NB: High dose ICS defined according to GINA
* One documented blood EOS (%) or absolute count in the last 12 months
* Twelve months of documented baseline data in medical records or asked on study visit day including asthma medication, especially oral corticosteroid (OCS) treatment and history of asthma exacerbations (number and severity)
* Evidence of one pre-bronchodilator forced expiratory volume in the first second (FEV1) in last 12 months or on study visit day
* Patients must be able and willing to read and comprehend written instructions, and comprehend and complete the questionnaires required by the protocol
* After full explanation, patients must have signed an informed consent document indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Other respiratory conditions including: chronic obstructive pulmonary disease (as main diagnosis), bronchiectasis, idiopathic pulmonary fibrosis, pulmonary hypertension, alpha-1-antitrypsine-deficiency, and malignancy of any kind (NB: the following conditions are permitted: nasal polyposis, allergic rhinitis, atopic dermatitis, non-idiopathic pulmonary fibrosis).
* Concurrent biologics for asthma except for stable allergen immunotherapy (defined as a stable dose and regimen at the time of the study visit). Acceptable washout periods for other asthma biologics:

  1. Other eosinophil lowering products indicated for asthma (including mepolizumab or reslizumab): at least 4 months.
  2. Prior omalizumab use: at least 1 month
* An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to complete questionnaires or participate in this study or impact the interpretations of results
* Patient is participating in an ongoing randomized clinical trial or participation in an observational trial that might, in the investigator's opinion, influence the assessment for the current study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged ≥ 18 years treated in primary or secondary care settings with diagnosed asthma defined as severe according American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines (iii).
Sampling Method: Non-Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Age at diagnosis | 1 year
  Age at diagnosis of asthma
Gender | 1 year
  Patient´s sex:
  Male Female
Ethnicity | 1 year
  Patient´s ethnic origin:
  White Black or African American Asian Other
Employment status | 1 year
  employed: full time/part time unemployed
Smoking status | 1 year
  Never former smoker current smoker
Blood eosinophiles (EOS) | 1 year
  % cells/microL
Immunoglobulin E (IgE) count | 1 year
  IU/ml
Fractional exhaled nitric oxide | 1 year
  ppb
Asthma medication | 1 year
  maintenance therapy
Chronic oral corticosteroids (OCS) use | 1 year
  Chronic OCS use (defined as treatment maintenance with OCS for ≥50% of the previous year) dose, start / stop, frequency
Short course systemic corticosteroids use | 1 year
  Short courses of systemic corticosteroids (or a temporary increase in a stable OCS background dose) for at least 3 days; a single depo-injectable dose of corticosteroids will be considered equivalent to a 3-day course of systemic corticosteroids dose, start / stop, frequency
Pre-bronchodilator FEV1 | 1 year
  Pre-bronchodilator FEV1
Asthma exacerbations | 1 year
  number severity (use of systemic inhaled corticosteroids (ICS); emergency department; inpatient hospital stay)
Healthcare resource use | 1 year
  number of visits to General Practitioner (GP), emergency room visits, hospitalizations, due to asthma
Charlson Comorbidity Index | 1 year
  Charlson Score calculated from yes/no answers to 19 questions on comorbidities and age.
  Comorbidity index range = 0-37 points; Age risk range = 0-5 points; Total Index range = 0-42 points 10-years-survival rate = 0-98% The higher the points, the higher the risk and the lower the 10-years-survival rate.
St George's Respiratory Questionnaire (SGRQ) | 4 weeks
  Health related quality of life questionnaire for patients with respiratory diseases.
  Subscales for "disease symptoms" , "activity", and "impact" . Each subscale can be calculated separately.
  The higher the score, the more severe the disease. A total score of all scales gives a measure for the total impact of the disease, range 0-100%.
Asthma Control Questionnaire (ACQ-6) | 4 weeks
  Level of asthma control as perceived by the patient. 6 questions with 6 predefined answers. Total points range 0 - 36. The higher, the worse the asthma control.
Medication adherence | 1 year
  Investigator´s discretion: yes/no

SECONDARY OUTCOMES:
Number of enrolled patients with severe asthma reported by investigators to be eligible for biological therapy among all enrolled patients with severe asthma | 1 year
Comparison of age between eligible and non-eligible patients for biologic therapy | 1 year
  Age (years)
Comparison of gender between eligible and non-eligible patients for biologic therapy | 1 year
  Gender at study visit (male/female)
Comparison of ethnicity between eligible and non-eligible patients for biologic therapy | 1 year
  Ethnicity ( White ,Black or African American, Asian , Other )
Comparison of socio-economic status between eligible and non-eligible patients for biologic therapy | 1 year
  Socio-economic status (employed/non employed)
Comparison of smoking history between eligible and non-eligible patients for biologic therapy | 1 year
  Smoking history (Former, current, Never smoker)
Comparison of blood eosinophiles between eligible and non-eligible patients for biologic therapy | 1 year
  Blood EOS (%) or (cells/microL)
Comparison of IgE counts between eligible and non-eligible patients for biologic therapy | 1 year
  IgE count (IU/L)
Comparison of fractional exhaled nitric oxide between eligible and non-eligible patients for biologic therapy | 1 year
  Fractional exhaled nitric oxide (FeNO)
Comparison of type of asthma medications for maintenance between eligible and non-eligible patients for biologic therapy | 1 year
  Asthma medications (type of maintenance therapies)
Comparison of type of oral corticosteroid use between eligible and non-eligible patients for biologic therapy | 1 year
  Chronic OCS use (defined as treatment maintenance with OCS for ≥50% of the previous year) or short courses of systemic corticosteroids (or a temporary increase in a stable OCS background dose) for at least 3 days; a single depo-injectable dose of corticosteroids will be considered equivalent to a 3-day course of systemic corticosteroids.
Comparison of pre-bronchodilator FEV1 between eligible and non-eligible patients for biologic therapy | 1 year
  Pre-bronchodilator FEV1 (L/sec)
Comparison of type of exacerbations between eligible and non-eligible patients for biologic therapy | 1 year
  Type of exacerbations (systemic steroids/ emergency department/ inpatient hospital stay)
Comparison of type of healthcare ressource use between eligible and non-eligible patients for biologic therapy | 1 year
  Healthcare ressource use (number of visits to GP, emergency room visits, hospitalisations, due to asthma)
Evaluation of age dependent on chronic OCS treatment or not | 1 year
  Age (years)
Evaluation of gender dependent on chronic OCS treatment or not | 1 year
  Gender at study visit (male/female)
Evaluation of ethnicity dependent on chronic OCS treatment or not | 1 year
  Ethnicity ( White ,Black or African American, Asian , Other )
Evaluation of socio-economic status dependent on chronic OCS treatment or not | 1 year
  Socio-economic status (employed/non employed)
Evaluation of smoking history dependent on chronic OCS treatment or not | 1 year
  Smoking history (Former, current, Never smoker)
Evaluation of blood eosinophiles dependent on chronic OCS treatment or not | 1 year
  Blood EOS (%) or (cells/microL)
Evaluation of IgE counts dependent on chronic OCS treatment or not | 1 year
  IgE count (IU/L)
Evaluation of fractional exhaled nitric oxide dependent on chronic OCS treatment or not | 1 year
  Fractional exhaled nitric oxide (FeNO)
Evaluation of asthma medications for maintenance dependent on chronic OCS treatment or not | 1 year
  Asthma medications (maintenance therapies)
Evaluation of pre-bronchodilato FEV1 dependent on chronic OCS treatment or not | 1 year
  Pre-bronchodilator FEV1 (L/sec)
Evaluation of type of exacerbations dependent on chronic OCS treatment or not | 1 year
  Type of exacerbations (systemic steroids/ emergency department/ inpatient hospital stay)
Evaluation of healthcare ressource use dependent on chronic OCS treatment or not | 1 year
  Healthcare resosurce use (number of visits to GP, emergency room visits, hospitalisations, due to asthma)
Reliability of physician´s assessment on eligibility for biologic therapy referral | 1 year
  Physician´s assessment on eligibility for biologic therapy referral: true/false

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Beier, MD, Principal Investigator — Deutsche Gesellschaft für Pneumologie
Locations (12):
- Research Site, Pleven, Bulgaria
- Research Site, Havířov, Czechia
- Research Site, Cappelle-en-Pévèle, Hauts-de-France, France
- Research Site, Reinfeld, Germany
- Research Site, Athens, Aigaleo, Greece
- Research Site, Budapest, Hungary
- Research Site, Sardinia, Sassari, Italy
- Research Site, Groningen, Netherlands
- Research Site, Wieruszów, Poland
- Research Site, Bacau, Romania
- Research Site, Slovenj Gradec, Slovenia
- Research Site, Málaga, Andalusia, Spain

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00039&attachmentIdentifier=293b0214-76ca-421f-b70b-1241835663c1&fileName=RECOGNISE_OS_report_synopsis_v1.0_2021-02-08_FINAL.pdf&versionIdentifier=